CLINICAL TRIAL: NCT06970210
Title: United4Stroke (U4S) - El Paso Network: Community Health Program With Group-Based Education
Brief Title: United4Stroke (U4S) - El Paso Network Stroke Community Program
Acronym: U4S
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas, El Paso (Other)
Responsible Party: Principal Investigator, Camila Torriani Pasin, Associate Professor, University of Texas, El Paso
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB#2153765
Record Dates: First submitted 2025-04-21; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-04

CONDITIONS: Stroke
Keywords: Stroke; Quality of Life; Sedentary Behaviors; Sedentary Lifestyle; Physical Inactivity; Community Health Education
MeSH Terms: conditions — Stroke; Sedentary Behavior; Health Education

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group-Based Education Only (Active Comparator): Participants assigned to the group-based education arm will attend the U4S program which will consist of group-based educational sessions led by research staff, covering topics such as physical activity, sedentary behavior, balance and fall prevention, and activities of daily living. This group will not receive individualized coaching aimed at increasing daily step count, but will receive a Fitbit to be worn during the program.
  Interventions: Behavioral: Group-Based Education
- Group-Based Education plus Individualized Coaching (Experimental): Participants assigned to the group-based education arm will attend the U4S program which will consist of group-based educational sessions led by research staff, covering topics such as physical activity, sedentary behavior, balance and fall prevention, and activities of daily living. This group will receive individualized coaching aimed at increasing daily step count, reducing sedentary behavior, and engaging in physical activities. They will also receive a Fitbit to be worn during the program.
  Interventions: Behavioral: Group-Based Education; Behavioral: Individualized Coaching

INTERVENTIONS:
Behavioral: Group-Based Education — The group-based education will consist of group sessions led by research staff, covering topics such as physical activity, sedentary behavior, balance and fall prevention, and activities of daily living. Social interactions amongst group members will be facilitated through group activities and discussions regarding the topics being discussed.
Behavioral: Individualized Coaching — Individualized coaching aims to increase the participants daily step count. Participants will be encouraged to achieve step count increases of 2%, 5%, or 10% per week or visit, depending on their readiness and willingness to progress. SMART goal-setting strategies will be employed to assist with the goal setting. Participants may also receive coaching related to reducing sedentary behavior and engaging in physical activities.
  Arms: Group-Based Education plus Individualized Coaching

SUMMARY:
What is United4Stroke (U4S)? United4Stroke is a research program at the University of Texas at El Paso (UTEP) that aims to help stroke survivors become more active and reduce sedentary time through education, movement, and personalized coaching.

Where Does It Happen?

All sessions take place at:

UTEP's Rehabilitation Sciences Complex located at 3333 North Mesa Street, El Paso, TX 79902

What is Involved?

The program includes 12 total visits over several months:

* 8 group sessions (held every two weeks)
* 4 individual evaluation visits (before, during, and after the program)

Who Can Participate?

* Individuals 18 years of age or older who have had a stroke at least 6 months prior to joining the study.
* Family caregivers may also join

What Happens During the Visits?

First Visit:

* Learn about the study and give consent
* Answer questions about memory, movement, general health, and daily activity
* Do walking and mobility tests
* Get fitted with a small movement sensor (ActivPAL) and a Fitbit

Group Sessions (Visits 2-8):

* Topics: physical activity, sitting less, balance and falls, and activities of daily living
* Led by UTEP physical therapy faculty
* Includes group discussions and hands-on activities
* Some participants will also get one-on-one coaching to help with physical activity engagement, daily step count, and reducing sedentary behavior.

Follow-Up Visits (Visits 9 and 11):

* Repeat earlier tests to check progress
* Share feedback about the program

Final Visit (Visit 10):

* Celebrate progress!
* Social gathering, certificates, and a presentation of results

Goal:

To support stroke survivors in becoming more active and living healthier, more independent lives-step by step.

DETAILED DESCRIPTION:
Specific Aims:

Aim 1: To evaluate the adherence rate, attendance, and satisfaction associated with a community health program that combines group-based education with individual coaching sessions for stroke survivors and their caregivers.

Hypothesis 1.1: A community health program incorporating group-based education and individual coaching sessions for stroke survivors will demonstrate acceptable rates of adherence and attendance.

Hypothesis 1.2: Stroke survivors and their caregivers will report satisfaction with a group-based education community health program.

Aim 2: To examine the effects of a community health program that combines group-based education with individual coaching sessions for stroke survivors and their caregivers on physical activity (PA), sedentary behavior (SB), and quality of life (QoL).

Hypothesis 2.1: The community health program, integrating group-based education with individual coaching sessions, will increase daily step count among stroke survivors more effectively than group-based education alone.

Hypothesis 2.2: The community health program, which combines group-based education with individual coaching sessions, will decrease SB among stroke survivors more effectively than group-based education alone.

Hypothesis 2.3: The community health program, which combines group-based education with individual coaching sessions, will improve the QoL of stroke survivors and their caregivers more effectively than group-based education alone.

Hypothesis 2.4: The one-month follow-up will show higher retention rates for the group intervention. Specifically, the community health program that combines group-based education with individual coaching will result in a greater rate of maintenance of daily step count, lower time spent in SB, and greater self-reported QoL one month after the program concludes when compared to group-based education alone.

Study Design and Methods:

The U4S project will employ a randomized controlled trial (RCT), following the Consolidated Standards of Reporting Trials (CONSORT) design. Participants will be recruited from community health centers and rehabilitation facilities throughout the Paso Del Norte region, supported by local healthcare providers and community organizations. A community engagement strategy will rely on ambassadors utilizing the partner mobile IT platform (High Enroll/ Patient Enroll) to promote the study through tailored marketing campaigns. Inclusion criteria are designed to ensure a focus on chronic stroke survivors: individuals aged 18 or older who are at least six months post-stroke, with the ability to participate in group sessions and provide informed consent. Recruitment will be facilitated through outreach to stroke support groups, healthcare providers, and community organizations within the region.

Recruitment and Participants:

Power calculations suggest that the RCT with a 5% significance level and moderate effect size (Cohen's f=0.5) will maintain 80% power with n=17 observations per group and 90% power with n=23 per group. This implies that with at least 46 total participants, we can maintain a well-powered experiment (90%), and with only 34 total subjects, we will have a moderately powered experiment (80%). All power calculations were performed in R 17 using the pwr package18. Over the course of 3 years, we aim to recruit 46 participants, averaging 23 participants per group (control and experimental). Each semester (3 semesters in total) will consist of two cohorts of 4 participants for each group, all of whom will be randomly assigned to either the control or intervention group. Participants in the control group will attend group-based education sessions covering essential stroke recovery topics, including awareness of PA engagement, reduction of SB, performance of activities of daily living (ADLs), and balance and fall risk. Group discussions will encourage social engagement, aiming to foster a sense of community and support among participants. In addition to the group education sessions, participants in the intervention group will receive one-on-one coaching from trained health professionals to set personalized health goals, with a primary focus on increasing daily step count. Coaching sessions will use motivational interviewing techniques to address ambivalence and enhance readiness for behavior change. Individualized action plans will be developed, focusing on the creation of SMART goals to incrementally increase daily steps. Based on baseline data or data collected at each visit, participants will be encouraged to achieve step count increases of 2%, 5%, or 10% per week or visit, depending on their readiness and willingness to progress. The intervention will span 12 weeks, with each group attending twelve visits at two-week intervals. Each session will last approximately one hour and a half, combining interactive education, group discussions, and individualized goal setting. The intervention integrates physical and psychosocial barriers and facilitators with SDH-focused strategies that address barriers commonly faced by Hispanic/Latino stroke survivors.

Description of Work:

This research project will encompass twelve visits to UTEP's Physical Therapy and Movement Sciences Department, where our laboratory is located. The first visit to the clinic will include the collection of demographics, sample characterization using scores from the Montreal Cognitive Assessment (MoCa), the Charlson Comorbidity Index (CCI), and the Fugl-Meyer Assessment of Motor Recovery after Stroke (FMA). We will also administer questionnaires that assess physical activity using the Human Activity Profile (HAP), sedentary behavior using the Sedentary Behavior Questionnaire (SBQ), and quality of life using the Stroke Impact Scale (SIS 3.0). Then, we will conduct several functional assessments including the Timed-Up-and-Go (TUG) test, the Five Times Sit to Stand Test (FTSTS), and the Ten Meters Walk Test (10MWT) in a randomized order. At the end of the visit, we will place an ActivPAL sensor on the stroke survivor that will record their number of steps, number of sit to stand transitions, and sedentary behavior based on the amount of time spent in different postural positions (i.e., sitting, lying) for seven days as a baseline measurement prior to the program. Randomization will be performed using sealed, opaque envelopes and the participant will be allocated to the respective group. Then, the stroke survivor and their caregiver (if applicable) will attend a first session with group-based education and the experimental group will receive their first individualized coaching. Zoom calls for the individualized coaching will be scheduled as needed. The program will be composed of seven additional sessions with group-based education and the experimental group will receive personalized coaching regarding step count increase after each session. The group sessions will be led by the principal investigator, and other research personnel. During these sessions, social interactions amongst the stroke survivors and caregivers will be highly encouraged through group activities and conversations. Then, the experimental group of stroke survivors will receive personalized coaching from the research team. Through this individualized coaching, our aim is to support stroke survivors throughout the states of the Transtheoretical Model of Health Behavioral Change. To accomplish this, we will provide the stroke survivors with guided and tailored exercises, set SMART (specific, measurable, achievable, realistic, and timed) goals every two weeks, help the participants in forming long-lasting habits, identify barriers that may restrict the stroke survivors from participating in physical activity, and make proposals to reduce those barriers to implement a more active lifestyle. During the eighth visit, we will also place the ActivPAL sensors onto the participants which will monitor their sedentary behavior based on time spent in different postural positions (i.e., sitting, lying) for seven days. This will serve as a post-program measurement. Then, the stroke survivors and caregivers will be invited back to the lab individually (visit 9) where the stroke survivors will respond to questionnaires that assess physical activity (HAP), sedentary behavior (SBQ), and quality of life (SIS 3.0). Then, we will conduct several functional assessments including the TUG test, the FTSTS test, and the 10MWT that will be conducted in a randomized order. The TUG test will be conducted over three trials consisting of familiarization, self-selected speed, and fast speed. The 10MWT will be conducted over four randomized trials, consisting of two self-selected speed trials, and two fast speed trials. The FTSTS test will be conducted over three trials, in which the participant will be asked to complete each trial as fast as they can. The caregiver will be administered a questionnaire that assesses strain that they may or may not experience as a caregiver (MCSI). During this visit, both the stroke survivor and caregiver will be administered a survey to assess their satisfaction with the program. Then, participants will be invited for a closing event (10th visit) with additional social interactions, games, and distribution of certificates of completion. One month after the closing event, the participants and their caregivers (if applicable) will be invited back for a follow-up assessment comprised of two visits. The follow-up assessment will consist of identical questionnaires, functional assessments, and sensor placement as those described in previous individual visits.

Data Analysis:

Aim 1: The analysis of adherence rate, attendance frequency, and satisfaction will be accomplished by using descriptive statistics and data visuals, including a general reporting of the mean, minimum and maximum levels observed.

Aim 2: The program's effect on measures of QoL, SB, and PA levels will be analyzed by computing a paired t-test between pre- and post- scores that are generated from the questionnaires and assessments described above for control and intervention groups.

Expected Results:

In the short term, the U4S project is expected to yield measurable improvements in the adherence, attendance, and satisfaction rates of chronic stroke survivors and their caregivers participating in the community-based program. The combined group-based education and individual coaching intervention is anticipated to enhance physical activity, reduce sedentary behavior, and improve quality of life. Outreach efforts with a community engagement strategy will likely result in increased community-wide awareness and participation in the study, surpassing recruitment benchmarks from previous stroke studies. The strategic use of targeted marketing, mobile IT platforms, and Ambassadors will ensure effective engagement with underserved Hispanic/Latino populations in the Paso del Norte region. These short-term outcomes will provide actionable insights into the feasibility and immediate impact of the intervention and the effectiveness of the recruitment strategies. Over the long term, the U4S project is expected to establish a sustainable and scalable community-academic partnership model for addressing health disparities in the Paso del Norte region and beyond. The program's success will provide a foundation for advancing evidence-based, culturally tailored interventions to improve rehabilitation outcomes for chronic stroke survivors. The findings will contribute to the scientific understanding of community-engaged health programs and inform policies to reduce health disparities in underserved populations.

The data and insights generated from this project will provide the essential evidence to refine our research questions, methodologies, and hypotheses. The evidence from this project will validate our innovative intervention approach, confirming its feasibility and potential effectiveness in improving the quality of life, physical activity, and self-reported health outcomes for stroke survivors and their caregivers within the Hispanic/Latino community.

ELIGIBILITY:
Inclusion Criteria: Individuals will be included if they are ≥ 18-years old, have had a stroke at least 6 months prior to baseline assessment, have a means of transportation to the UTEP physical therapy building to attend the program/visits, and are clinically stable (the participant's health is not rapidly worsening and there may be a level of stability in their overall health status).

Exclusion Criteria: Individuals will be excluded if they are unable to consent, if they do not have a means of transportation to attend the program/study visits, if they require a caregiver and the caregiver is unable to attend, if they walk greater than an average of 7,000 steps a day, if they walk at a speed less than or equal to 0.3 m/s, or if the participant attends less than 60% of the group-based educational sessions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-06-02 (Estimated); Primary Completion 2028-12-20 (Estimated); Study Completion 2028-12-20 (Estimated)

PRIMARY OUTCOMES:
Daily Step Count | Baseline, week 6 (during intervention), week 13 (post-intervention), and week 19 (follow-up).
  Daily step count data will be collected.

SECONDARY OUTCOMES:
Sedentary Behavior (Objective) | Baseline, week 6 (during intervention), week 13 (post-intervention), and week 19 (follow-up).
  Sedentary behavior will be assessed using the ActivPAL sensor, which will be adhered to the participant's thigh and worn continuously for seven days. The ActivPAL monitors posture and movement, providing detailed data on time spent sitting, standing, walking, and lying down. Additionally, the sensor provides data of daily sit to stand transition counts. Sensors will be deployed at four timepoints: baseline, mid-program, post-intervention, and follow-up.
Sedentary Behavior (Subjective) | Baseline, week 13 (post-intervention), and week 19 (follow-up).
  Data for sedentary behavior will be collected using the Sedentary Behavior Questionnaire (SBQ). This questionnaire asked the participants how long they believe they spend participating in 11 different activities during week and weekend days.
Quality of Life (QoL) | Baseline, week 13 (post-intervention), and week 19 (follow-up).
  Data on QoL will be collected using the Stroke Impact Scale (SIS 3.0). The Stroke Impact Scale (SIS) is a self-report questionnaire that evaluates disability and health-related quality of life after stroke (Mudler & Nijland, 2016). It is a 59-item questionnaire, assessing eight domains: strength, hand function, activities of daily living, mobility, communication, emotion, memory and thinking, and participation/role function. Each item is presented as a 5-point Likert scale, allowing the participant to rate the level of difficulty they experience in completing each item. Additionally, the participant is asked to rate how much they think that they have recovered from their stroke on a 0-100 scale.
Quality of Life (QoL) | Baseline, week 13 (post-intervention), and week 19 (follow-up).
  Data on QoL will be collected using the Modified Caregiver Strain Index (MCSI). The MCSI is a 13 item questionnaire administered to caregivers (if applicable). The questionnaire assesses strain related to the following domains: financial, physical, psychological, social, and personal. Higher scores indicate more strain.
Mobility Performance | Baseline, week 13 (post-intervention), and week 19 (follow-up).
  Data for mobility performance will be collected using the Timed-Up-and-Go Test (TUG). The TUG test assesses mobility and fall risk. During the test, the participant is instructed to stand up from a chair, walk three meters, turn around, walk back to the chair, and sit back down. The test will be conducted over three trials: familiarization, self-selected speed, and fast speed.
Mobility Performance | Baseline, week 13 (post-intervention), and week 19 (follow-up).
  Data for mobility performance will be collected using the Five Times Sit to Stand (FTSTS) Test. The FTSTS test assesses functional mobility and strength. During the test, the participant is instructed to rise to a full standing position and return to sitting five times as quickly as possible, without using their arms.
Mobility Performance | Baseline, week 13 (post-intervention), and week 19 (follow-up).
  Data for mobility performance will be collected using the Ten Meters Walk Test (10MWT). The 10MWT assesses functional mobility and gait. During the test, the participant is instructed to walk 10 meters (with 2 additional meters on each end of the walkway for acceleration and deceleration). The test will be conducted over 4 trials presented in a randomized order: 2 self-selected comfortable walking speed, and 2 at a fast walking speed.

OTHER OUTCOMES:
Feasibility (adherence) | Weeks 1-14 (intervention period)
  Feasibility outcomes will be measured by adherence rate (number of participants invited to program compared to the number of participants who engaged in the program).
Feasibility (attendance frequency) | Weeks 1-14 (intervention period)
  Feasibility outcomes will be measured by attendance frequency (total number of sessions that each participant attended).
Feasibility (satisfaction) | Week 13 (post-intervention)
  Feasibility outcomes will be measured by participant satisfaction (Likert-scale questionnaire administered after completion of the program).

CONTACTS AND LOCATIONS:
Overall Officials: Camila Torriani-Pasin, PhD, PT, Principal Investigator — The University of Texas at El Paso
Locations (1):
- The University of Texas at El Paso: Rehabilitation Sciences Complex, El Paso, Texas, United States

IPD SHARING:
Plan to Share IPD: No
While we recognize the value of data sharing in advancing scientific knowledge, we have chosen not to share individual participant data (IPD) from this study due to ethical and logistical considerations. This study involves a vulnerable population (stroke survivors and potentially their caregivers), and the dataset includes sensitive health information that, even when de-identified, may pose a risk of re-identification given the relatively small sample size and the community-based nature of recruitment. Additionally, our informed consent process does not include provisions for broad data sharing, in order to respect participants' privacy and autonomy.
  Furthermore, at this stage, we lack the infrastructure necessary to ensure secure and ethical access to IPD for external researchers. Future data sharing may be considered upon appropriate ethical approval and with participant consent, aligned with best practices and institutional policies.

REFERENCES:
- [Background] Gladstone DJ, Danells CJ, Black SE. The fugl-meyer assessment of motor recovery after stroke: a critical review of its measurement properties. Neurorehabil Neural Repair. 2002 Sep;16(3):232-40. doi: 10.1177/154596802401105171. PMID 12234086
- [Background] Patrick H, Williams GC. Self-determination theory: its application to health behavior and complementarity with motivational interviewing. Int J Behav Nutr Phys Act. 2012 Mar 2;9:18. doi: 10.1186/1479-5868-9-18. PMID 22385676
- [Background] Hashemzadeh M, Rahimi A, Zare-Farashbandi F, Alavi-Naeini AM, Daei A. Transtheoretical Model of Health Behavioral Change: A Systematic Review. Iran J Nurs Midwifery Res. 2019 Mar-Apr;24(2):83-90. doi: 10.4103/ijnmr.IJNMR_94_17. PMID 30820217
- [Background] Thompson ED, Pohlig RT, McCartney KM, Hornby TG, Kasner SE, Raser-Schramm J, Miller AE, Henderson CE, Wright H, Wright T, Reisman DS. Increasing activity after stroke: a randomized controlled trial of highintensity walking and step activity intervention. medRxiv [Preprint]. 2023 Aug 9:2023.03.11.23287111. doi: 10.1101/2023.03.11.23287111. PMID 37609269
- [Background] Shumway-Cook A, Brauer S, Woollacott M. Predicting the probability for falls in community-dwelling older adults using the Timed Up & Go Test. Phys Ther. 2000 Sep;80(9):896-903. PMID 10960937
- [Background] Thornton M, Travis SS. Analysis of the reliability of the modified caregiver strain index. J Gerontol B Psychol Sci Soc Sci. 2003 Mar;58(2):S127-32. doi: 10.1093/geronb/58.2.s127. PMID 12646602
- [Background] Ruescas-Nicolau MA, Sanchez-Sanchez ML, Cortes-Amador S, Perez-Alenda S, Arnal-Gomez A, Climent-Toledo A, Carrasco JJ. Validity of the International Physical Activity Questionnaire Long Form for Assessing Physical Activity and Sedentary Behavior in Subjects with Chronic Stroke. Int J Environ Res Public Health. 2021 Apr 29;18(9):4729. doi: 10.3390/ijerph18094729. PMID 33946690
- [Background] O'Keefe LM, Doran SJ, Mwilambwe-Tshilobo L, Conti LH, Venna VR, McCullough LD. Social isolation after stroke leads to depressive-like behavior and decreased BDNF levels in mice. Behav Brain Res. 2014 Mar 1;260:162-70. doi: 10.1016/j.bbr.2013.10.047. Epub 2013 Nov 5. PMID 24211537
- [Background] Moher D, Hopewell S, Schulz KF, Montori V, Gotzsche PC, Devereaux PJ, Elbourne D, Egger M, Altman DG. CONSORT 2010 explanation and elaboration: updated guidelines for reporting parallel group randomised trials. BMJ. 2010 Mar 23;340:c869. doi: 10.1136/bmj.c869. No abstract available. PMID 20332511
- [Background] Cheng DK, Nelson M, Brooks D, Salbach NM. Validation of stroke-specific protocols for the 10-meter walk test and 6-minute walk test conducted using 15-meter and 30-meter walkways. Top Stroke Rehabil. 2020 May;27(4):251-261. doi: 10.1080/10749357.2019.1691815. Epub 2019 Nov 21. PMID 31752634
- [Background] Bailey RR. Goal Setting and Action Planning for Health Behavior Change. Am J Lifestyle Med. 2017 Sep 13;13(6):615-618. doi: 10.1177/1559827617729634. eCollection 2019 Nov-Dec. PMID 31662729
- [Background] Lang CE, Holleran CL, Strube MJ, Ellis TD, Newman CA, Fahey M, DeAngelis TR, Nordahl TJ, Reisman DS, Earhart GM, Lohse KR, Bland MD. Improvement in the Capacity for Activity Versus Improvement in Performance of Activity in Daily Life During Outpatient Rehabilitation. J Neurol Phys Ther. 2023 Jan 1;47(1):16-25. doi: 10.1097/NPT.0000000000000413. Epub 2022 Aug 4. PMID 35930404
- [Background] Robinson BC. Validation of a Caregiver Strain Index. J Gerontol. 1983 May;38(3):344-8. doi: 10.1093/geronj/38.3.344. PMID 6841931
- [Background] Vellone E, Savini S, Fida R, Dickson VV, Melkus GD, Carod-Artal FJ, Rocco G, Alvaro R. Psychometric evaluation of the Stroke Impact Scale 3.0. J Cardiovasc Nurs. 2015 May-Jun;30(3):229-41. doi: 10.1097/JCN.0000000000000145. PMID 24695074
- [Background] Ezzati A, Jiang J, Katz MJ, Sliwinski MJ, Zimmerman ME, Lipton RB. Validation of the Perceived Stress Scale in a community sample of older adults. Int J Geriatr Psychiatry. 2014 Jun;29(6):645-52. doi: 10.1002/gps.4049. Epub 2013 Dec 3. PMID 24302253
- [Background] Rosenberg DE, Norman GJ, Wagner N, Patrick K, Calfas KJ, Sallis JF. Reliability and validity of the Sedentary Behavior Questionnaire (SBQ) for adults. J Phys Act Health. 2010 Nov;7(6):697-705. doi: 10.1123/jpah.7.6.697. PMID 21088299
- [Background] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Background] Teixeira-Salmela LF, Devaraj R, Olney SJ. Validation of the human activity profile in stroke: a comparison of observed, proxy and self-reported scores. Disabil Rehabil. 2007 Oct 15;29(19):1518-24. doi: 10.1080/09638280601055733. PMID 17852225
- [Background] Wei X, Ma Y, Wu T, Yang Y, Yuan Y, Qin J, Bu Z, Yan F, Zhang Z, Han L. Which cutoff value of the Montreal Cognitive Assessment should be used for post-stroke cognitive impairment? A systematic review and meta-analysis on diagnostic test accuracy. Int J Stroke. 2023 Oct;18(8):908-916. doi: 10.1177/17474930231178660. PMID 37190789
- [Background] Chiti G, Pantoni L. Use of Montreal Cognitive Assessment in patients with stroke. Stroke. 2014 Oct;45(10):3135-40. doi: 10.1161/STROKEAHA.114.004590. Epub 2014 Aug 12. No abstract available. PMID 25116881
- [Background] Carson N, Leach L, Murphy KJ. A re-examination of Montreal Cognitive Assessment (MoCA) cutoff scores. Int J Geriatr Psychiatry. 2018 Feb;33(2):379-388. doi: 10.1002/gps.4756. Epub 2017 Jul 21. PMID 28731508
- [Background] Weltermann BM, Homann J, Rogalewski A, Brach S, Voss S, Ringelstein EB. Stroke knowledge among stroke support group members. Stroke. 2000 Jun;31(6):1230-3. doi: 10.1161/01.str.31.6.1230. PMID 10835437
- [Background] Muller M, Toth-Cohen S, Mulcahey MJ. Development and evaluation of a hospital-based peer support group for younger individuals with stroke. Occup Ther Health Care. 2014 Jul;28(3):277-95. doi: 10.3109/07380577.2014.919551. PMID 24971895
- [Background] Lin FH, Yih DN, Shih FM, Chu CM. Effect of social support and health education on depression scale scores of chronic stroke patients. Medicine (Baltimore). 2019 Nov;98(44):e17667. doi: 10.1097/MD.0000000000017667. PMID 31689780
- [Background] Louie SW, Liu PK, Man DW. The effectiveness of a stroke education group on persons with stroke and their caregivers. Int J Rehabil Res. 2006 Jun;29(2):123-9. doi: 10.1097/01.mrr.0000191851.03317.f0. PMID 16609323
- [Background] Christensen ER, Golden SL, Gesell SB. Perceived Benefits of Peer Support Groups for Stroke Survivors and Caregivers in Rural North Carolina. N C Med J. 2019 May-Jun;80(3):143-148. doi: 10.18043/ncm.80.3.143. PMID 31072940
- [Background] U.S. Census Bureau Quickfacts: El Paso City, Texas. United States Bureau Census . (n.d.). https://www.census.gov/quickfacts/fact/table/elpasocitytexas/POP01022
- [Background] Hernandez R, Carnethon M, Giachello AL, Penedo FJ, Wu D, Birnbaum-Weitzman O, Giacinto RE, Gallo LC, Isasi CR, Schneiderman N, Teng Y, Zeng D, Daviglus ML. Structural social support and cardiovascular disease risk factors in Hispanic/Latino adults with diabetes: results from the Hispanic Community Health Study/Study of Latinos (HCHS/SOL). Ethn Health. 2018 Oct;23(7):737-751. doi: 10.1080/13557858.2017.1294660. Epub 2017 Feb 23. PMID 28277024
- [Background] Chambers EC, Hanna DB, Hua S, Duncan DT, Camacho-Rivera M, Zenk SN, McCurley JL, Perreira K, Gellman MD, Gallo LC. Relationship between area mortgage foreclosures, homeownership, and cardiovascular disease risk factors: The Hispanic Community Health Study/Study of Latinos. BMC Public Health. 2019 Jan 17;19(1):77. doi: 10.1186/s12889-019-6412-2. PMID 30654781
- [Background] Trifan G, Gallo LC, Lamar M, Garcia-Bedoya O, Perreira KM, Pirzada A, Talavera GA, Smoller SW, Isasi CR, Cai J, Daviglus ML, Testai FD. Association of Unfavorable Social Determinants of Health With Stroke/Transient Ischemic Attack and Vascular Risk Factors in Hispanic/Latino Adults: Results From Hispanic Community Health Study/Study of Latinos. J Stroke. 2023 Sep;25(3):361-370. doi: 10.5853/jos.2023.00626. Epub 2023 Aug 10. PMID 37554075
- [Background] Northcott S, Moss B, Harrison K, Hilari K. A systematic review of the impact of stroke on social support and social networks: associated factors and patterns of change. Clin Rehabil. 2016 Aug;30(8):811-31. doi: 10.1177/0269215515602136. Epub 2015 Sep 1. PMID 26330297
- [Background] House JS, Landis KR, Umberson D. Social relationships and health. Science. 1988 Jul 29;241(4865):540-5. doi: 10.1126/science.3399889.
- [Background] Berkman LF. The relationship of social networks and social support to morbidity and mortality. In: Cohen SS, ed. Social support and health. New York: Academic Press, 1985;240-259.
- [Background] Brummett BH, Barefoot JC, Siegler IC, Clapp-Channing NE, Lytle BL, Bosworth HB, Williams RB Jr, Mark DB. Characteristics of socially isolated patients with coronary artery disease who are at elevated risk for mortality. Psychosom Med. 2001 Mar-Apr;63(2):267-72. doi: 10.1097/00006842-200103000-00010. PMID 11292274
- [Background] Michael YL, Colditz GA, Coakley E, Kawachi I. Health behaviors, social networks, and healthy aging: cross-sectional evidence from the Nurses' Health Study. Qual Life Res. 1999 Dec;8(8):711-22. doi: 10.1023/a:1008949428041. PMID 10855345
- [Background] Vogt TM, Mullooly JP, Ernst D, Pope CR, Hollis JF. Social networks as predictors of ischemic heart disease, cancer, stroke and hypertension: incidence, survival and mortality. J Clin Epidemiol. 1992 Jun;45(6):659-66. doi: 10.1016/0895-4356(92)90138-d. PMID 1607905
- [Background] Knox SS, Siegmund KD, Weidner G, Ellison RC, Adelman A, Paton C. Hostility, social support, and coronary heart disease in the National Heart, Lung, and Blood Institute Family Heart Study. Am J Cardiol. 1998 Nov 15;82(10):1192-6. doi: 10.1016/s0002-9149(98)00599-2. PMID 9832093
- [Background] Boden-Albala B, Litwak E, Elkind MS, Rundek T, Sacco RL. Social isolation and outcomes post stroke. Neurology. 2005 Jun 14;64(11):1888-92. doi: 10.1212/01.WNL.0000163510.79351.AF. PMID 15955939
- [Background] Feigin VL, Brainin M, Norrving B, Martins S, Sacco RL, Hacke W, Fisher M, Pandian J, Lindsay P. World Stroke Organization (WSO): Global Stroke Fact Sheet 2022. Int J Stroke. 2022 Jan;17(1):18-29. doi: 10.1177/17474930211065917. PMID 34986727
- [Background] GBD 2019 Stroke Collaborators. Global, regional, and national burden of stroke and its risk factors, 1990-2019: a systematic analysis for the Global Burden of Disease Study 2019. Lancet Neurol. 2021 Oct;20(10):795-820. doi: 10.1016/S1474-4422(21)00252-0. Epub 2021 Sep 3. PMID 34487721